CLINICAL TRIAL: NCT04103814
Title: Effect of Topical CBD Oil on Pain Scores for Hallux Disorders: A Randomized Controlled Trial
Brief Title: Effect of Topical CBD Cream for Degenerative Hallux Disorders
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of resources to continue enrollment
Sponsor: Rush University Medical Center (Other)
Collaborators: Mid-America Orthopaedic Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19052902
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Hallux Valgus; Hallux Rigidus
MeSH Terms: conditions — Hallux Valgus; Hallux Rigidus

STUDY DESIGN:
Intervention Model Description: Enrolled patients will receive either active Mg-CBDa (magnesium-cannabidiolic acid) cream or placebo cream (neutral emollient containing no active agent) for topical treatment of hallux rigidus or hallux valgus.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mg-CBDa cream (Active Comparator): Subjects in this group will receive the active Mg-CBDa (magnesium-cannabidiolic acid) for topical treatment of hallux valgus or hallux rigidus.
  Interventions: Drug: magnesium-cannabidiolic acid cream
- Placebo cream (Placebo Comparator): Subjects in this group will receive the inactive CBD cream for topical treatment of hallux valgus or hallux rigidus. The ingredients of the placebo cream are: butyrospermum parkii (shea butter), caprylic/capric triglycerides medium-chain triglycerides (MCT oil), and food coloring to match the CBD oil. There will be 345 grams of shea butter and 62ml MCT oil per batch.
  Interventions: Drug: Placebo cream

INTERVENTIONS:
Drug: magnesium-cannabidiolic acid cream — Patients will receive Mg-CBDa (magnesium-cannabidiolic acid) cream for topical treatment of hallux rigidus or hallux valgus.
  Arms: Mg-CBDa cream
Drug: Placebo cream — Patients will receive placebo cream (neutral emollient containing no active agent) for topical treatment of hallux rigidus or hallux valgus. The ingredients of the placebo cream are as follows: Butyrospermum parkii (shea butter), caprylic/capric triglycerides medium-chain triglycerides (MCT oil), food coloring to match the CBD oil. There will be 345 grams of shea butter and 62ml MCT oil per batch.
  Arms: Placebo cream

SUMMARY:
Hallux rigidus and hallux valgus are chronic forefoot conditions associated with pain, inflammation and functional impairment. Topical cannabidiol (CBD) cream has been shown to decrease inflammation, swelling, and pain response in arthritis models with minimal side effects, although the intervention has never been studied in hallux valgus or hallux rigidus. The purpose of this study is to determine if topical CBD cream is an effective treatment for pain secondary to hallux rigidus and hallux valgus.

DETAILED DESCRIPTION:
Hallux rigidus and hallux valgus are chronic forefoot conditions associated with pain, inflammation and functional impairment. While operative interventions exist, nonoperative modalities are the mainstay of treatment for most patients. Options include shoe wear modification, manual and physical therapy, intraarticular injection of corticosteroids or sodium hyaluronate, oral nonsteroidal anti-inflammatories, and foot orthoses. Oral anti-inflammatories are the most effective non-operative strategy, but unfortunately, are associated with major adverse side effects and are contraindicated in many patients. Topical cannabidiol (CBD) cream has been shown to decrease inflammation, swelling, and pain response in arthritis models with minimal side effects, although the intervention has never been studied in hallux valgus or hallux rigidus. This prospective randomized trial will compare topical CBD cream vs placebo cream for the treatment of pain secondary to hallux valgus and hallux rigidus. The primary outcome of interest in the change in pre and post-treatment Visual Analog System (VAS) pain scores. VAS pain score is a measurement on a continuum of values of pain intensity. The purpose of this study is to determine if topical CBD cream is an effective treatment for pain secondary to hallux rigidus and hallux valgus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a new diagnosis of hallux rigidus or hallux valgus
* VAS pain score of 4 or higher
* Age > 18 years
* The patient provides informed consent

Exclusion Criteria:

* A previous operative procedure to the first metatarsal for treatment of hallux valgus or hallux rigidus
* VAS pain score at presentation less than 4
* Concomitant hallux valgus and hallux rigidus on the ipsilateral side
* Allergy to CBD, Cannabidiolic acid (CBDa) or any other ingredient contained in the topical cream
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-10-20 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Lee, MD, Principal Investigator — Midwest Orthopaedics at Rush
Locations (1):
- Midwest Orthopaedics at Rush, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CBD Cream: Patients will be treated with CBD cream
- Control: Patients will be treated with a placebo cream not containing CBD
Period: Overall Study
Arm/Group | CBD Cream | Control
Started | 8 | 3
Completed | 0 | 0
Not Completed | 8 | 3

BASELINE CHARACTERISTICS:
Population: study terminated as it was too resource intensive to obtain pain scores from patients
Groups:
- CBD Cream: Patients will be randomized to CBD cream
- Control: Patients will be randomized to a placebo cream without CBD
- Total: Total of all reporting groups
Arm/Group | CBD Cream | Control | Total
Number analyzed (Participants) | 8 | 3 | 11
Age, Categorical [Count of Participants; unit: Participants] — No data was collected Population: No data were collected/analyzed
Age, Continuous [Mean (Standard Deviation); unit: years] — No data was collected or analyzed. Population: study terminated as it was too resource-intensive to obtain pain scores from patients as a result, no data was collected or analyzed.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: No data were collected/analyzed.
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: No data were collected/analyzed
Region of Enrollment [Number; unit: participants]
  United States | 8 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Post-treatment VAS Score Averaged Daily Over 4 Weeks.
Description: Weekly visual analog system (VAS) pain scores will be measured daily for four weeks. The VAS pain score is a measure of pain severity. It is measured on a scale from 0 to 10, with 10 being the worst pain the patient has experienced. No patients completed full enrollment so no data was analyzed.
Time Frame: 4 weeks
Population: No data were analyzed for this outcome because there were no participants data collected.
Groups:
- CBD Cream vs Placebo: Patients will be randomized to CBD cream vs Placebo
Arm/Group | CBD Cream vs Placebo
Number analyzed (Participants) | 0

2. Primary Outcome: Weekly Foot Function Index
Description: The foot function index (FFI) is a questionnaire that measures foot pain and disability. It is self-administered and consists of 23 items divided into 3 subscales (pain, disability, and activity limitation). The pain subcategory consists of 9 questions (scored out of 90) and is a measure of pain in different situations, such as walking with shoes versus barefoot. The disability subcategory consists of 9 questions (scored out of 90) and measures functional activities, such as difficulty walking upstairs. The activity limitation subcategory consists of 5 questions (scored out of 50) and measures limitations caused by the foot problem. All three subcategories are summed together to get a final number, with higher numbers indicating worse pain.
Time Frame: 4 weeks
Population: No data were analyzed for this outcome because there were no participants data collected
Arm/Group | CBD Cream vs Placebo
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The time period of adverse event data was collected for 6 months
Arm/Group | Mg-CBDa Cream | Placebo Cream
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT04103814/Prot_000.pdf
  • Informed Consent Form (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT04103814/ICF_001.pdf